CLINICAL TRIAL: NCT03290534
Title: Feasibility Study to Treat Lung Cancer With the Permanently Implantable LDR CivaSheet®
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CivaTech Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT006
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer; Lung Cancer Stage I; Lung Cancer Stage II
Keywords: wedge resection; sublobar resection; brachytherapy; CivaSheet; Pd-103; CivaTech Oncology; lung cancer; lung
MeSH Terms: conditions — Lung Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CivaSheet Directional LDR Brachytherapy (Experimental): FDA Cleared CivaSheet directional Pd-103 Brachytherapy Source is a planar radiation source which utilizes gold shielding in its construction. This device is radioactive on one side only, and is capable of safely delivering high doses of radiation to target areas even when placed directly adjacent to sensitive, healthy tissue or critical structures.
  Interventions: Device: CivaSheet

INTERVENTIONS:
Device: CivaSheet — implanting CivaSheet for localized radiation dose delivery
  Other Names: brachytherapy

SUMMARY:
This is a feasibility study to determine the usefulness of a brachytherapy device that utilizes active components (palladium-103) of standard devices in a novel configuration, which may benefit lung cancer patients by reducing the radiation dose to critical structures, such as the heart wall, while giving a therapeutic dose to diseased tissue, such as at a surgical margin.

ELIGIBILITY:
Inclusion Criteria:

* Subject signed inform consent
* Suspected or proven non-small cell lung cancer (NSCLC) in the upper lobes of the left or right lung
* Pre-operative criteria
* Lung nodule suspicious for NSCLC
* Mass ≤ 7 cm in maximum diameter by CT scan of the chest and upper abdomen
* Clinical stage I or Clinical stage II
* Not pregnant or nursing
* Negative pregnancy test in premenopausal women
* Fertile patients must use effective contraception
* More than 5 years since prior invasive malignancy unless non melanoma skin cancer or in-situ cancer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Local Control Rate at 1 year | 1 year
  The local control rate in the region irradiated by CivaSheet.

SECONDARY OUTCOMES:
Freedom from regional or distant recurrence | 1 year
  Control rate for recurrences outside the local area irradiated by CivaSheet.
Time to recurrence | 1 year
  Time in months to any recurrence
Toxicity graded on CTCAE 4.0 Scale | 1 year
  pulmonary function, radiation pneumonitis, fatigue, lung fibrosis, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No